CLINICAL TRIAL: NCT07262190
Title: Implementing a Patient Navigation Intervention Across a Health System to Improve Outcomes for Patients With Opioid Use Disorder
Brief Title: NavSTAR Implementation Effectiveness Trial Across a Health System
Acronym: Philly NavSTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: Thomas Jefferson University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: R33DA059033 (NIH); R33DA059033 (NIH)
Record Dates: First submitted 2025-10-23; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
Keywords: patient navigation
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster randomized design will be used, in which all five sites begin in a control phase and are sequentially randomized to cross over to the intervention at staggered time points, permitting both within-site and between-site comparisons over time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Treatment as usual consists of standard management by the medical or surgical team during inpatient admission, and usual care from the addiction consult service, if applicable, which provides social work consults, withdrawal symptom management, and initiation of naltrexone, buprenorphine, or methadone. All standard hospital services will be available to participants.
- NavSTAR (Experimental): NavSTAR consists of TAU plus contact with a trained patient navigator who delivers the NavSTAR intervention, inclusive of theory-based motivational content, during and after discharge from the hospital. The patient navigator also has access to a small participant fund to assist with overcoming structural barriers to care (e.g., phone, obtaining IDs, a meal, a taxi ride etc.). Using the NavSTAR PN manual, the PN will address internal and external barriers to engagement in OAT through motivational intervention techniques and proactive case management and care coordination services. Contact with the PN begins at the bedside while the participant is admitted to the hospital and continues for 3 months after discharge
  Interventions: Behavioral: NavSTAR (Philly adaptation)

INTERVENTIONS:
Behavioral: NavSTAR (Philly adaptation) — NavSTAR consists of TAU plus contact with a trained patient navigator who delivers the NavSTAR intervention, inclusive of theory-based motivational content, during and after discharge from the hospital. The patient navigator also has access to a small participant fund to assist with overcoming structural barriers to care (e.g., phone, obtaining IDs, a meal, a taxi ride etc.). Using the NavSTAR PN manual, the PN will address internal and external barriers to engagement in OAT through motivational intervention techniques and proactive case management and care coordination services. Contact with the PN begins at the bedside while the participant is admitted to the hospital and continues for 3 months after discharge
  Arms: NavSTAR

SUMMARY:
Patient Navigation (PN) interventions following hospitalization can improve outcomes for people with opioid use disorder treatment. Delivering PN interventions on a wide scale requires many resources and coordination across institutions. This will use an evidence-based process to find solutions to these significant barriers by engaging community, hospital, and patient partners. This study is being conducted to learn more about how to implement NavSTAR, a patient navigation intervention for people with opioid use disorder, across a health system. The research team showed in a previous study with 400 participants that NavSTAR significantly increased entry into opioid use disorder treatment, reduced readmissions to the hospital, and was highly cost- effective compared to treatment as usual. This study will first pilot NavSTAR with 32 patient participants across 4 hospitals in the City of Philadelphia. Then, a large trial with 720 patient participants will be conducted to see if people who need the intervention are reached, and a sustainable plan will be created to continue the intervention after the grant award period.

DETAILED DESCRIPTION:
Opioid agonist treatment (OAT) is protective against overdose, yet less than 20% of people with opioid use disorder (OUD) engage in such treatment. Hospital utilization is high among people with OUD and can be a 'reachable moment' to initiate OAT. However, most hospitals lack the capacity to follow up with patients after discharge. Patient navigation (PN) interventions following hospital discharge can help patients engage in OAT and navigate complex systems of care. However, challenges persist in implementing PN interventions on a wide scale, as they require coordination across organizations, data sharing, dedicated personnel, and resources. To bring these interventions to scale, strategies are needed to determine feasibility, reach, and sustainability. Testing innovative implementation strategies for PN interventions has the potential for significant impact, as it will demonstrate implementation success of an intervention that can address the opioid epidemic in real-world settings and close the research-to-practice translation gap. The proposed study is a type II hybrid implementation-effectiveness trial of Navigation Services to Avoid Rehospitalization (NavSTAR). The research team showed in a single-site randomized trial with 400 participants that NavSTAR significantly improved OAT entry, reduced readmissions, and was highly cost-effective compared to treatment as usual. The present study will test an Implementation Facilitation (IF) strategy to provide training, resources, and performance feedback to implement NavSTAR in five hospitals in Philadelphia. It is hypothesized that engaging stakeholders in an IF strategy will yield an implementation process that is feasible, acceptable, and effective in improving outcomes for patients with OUD. During the R33 phase, a type II hybrid-implementation-effectiveness trial of NavSTAR will be conducted with 720 participants using a randomized stepped-wedge design.

The proposed study is a type II hybrid implementation-effectiveness trial of Navigation Services to Avoid Rehospitalization (NavSTAR). The present study will test an Implementation Facilitation (IF) strategy following Proctor's conceptual model of implementation, using an external facilitator and internal local clinical champions to provide training, resources and performance feedback to implement NavSTAR in five hospitals. It is hypothesized that engaging stakeholders in an IF strategy will yield an implementation process that is feasible, acceptable, and effective in expanding engagement in OAT post-discharge. This type II hybrid implementation-effectiveness randomized stepped-wedge trial (N=720) will examine NavSTAR's sustained use in a hospital system to improve outcomes for patients with OUD.

R33 Specific Aims:

* Aim 1: Determine the successful implementation of NavSTAR in terms of a) feasibility, b) reach, and c) sustainability using the newly developed hospital system protocol.
* Aim 2: Determine the effectiveness of NavSTAR to a) improve OAT initiation in the three months post-discharge, b) decrease hospital utilization (inpatient readmissions and emergency department visits), c) reduce overdoses (fatal and non-fatal), and d) improve other patient outcomes (e.g., quality of life, substance use).

The proposed study has high public health significance because it will develop and test an implementation strategy for an intervention (NavSTAR) to improve OAT engagement and outcomes for patients with OUD. The study will yield novel data on how best to implement NavSTAR across a health system operating in an epicenter of the OUD crisis. Study findings will help to develop a path to scale-up this important intervention to address the opioid epidemic.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older;
2. current DSM-5 criteria for moderate to severe OUD;
3. willing and able to provide informed consent in English.

Exclusion Criteria:

1. enrollment in OUD treatment 30-days prior to hospitalization;
2. residency outside the City of Philadelphia;
3. pregnancy;
4. planned discharge to a long-term inpatient care facility (e.g., hospice);
5. hospitalization for a suicide attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Opioid Agonist Treatment initiation | 3 months
  Post-discharge rate of OAT initiation will be ascertained via health record review and self-report with verification through records where applicable (e.g., Community Behavioral Health system).

SECONDARY OUTCOMES:
Feasibility: Demonstrated ability to enroll participants in the intervention | From baseline until end of study, approximately 30 months
  Feasibility will be measured based on the number of participants who received the intervention during the implementation period.
Inpatient readmissions (30 days) | 30 days
  Information on acute care hospital inpatient readmission within 30 days will be assessed using health records and self-report (in the event of inconsistency, objective data will dominate).
Inpatient readmissions | through 3, 6, and 12 months
  Inpatient hospital readmissions (number of events) will be assessed using health record review and self-report (in the event of inconsistencies, objective data will dominate).
Emergency department visits | through 3, 6, and 12 months
  Emergency Department utilization (number of events) will be assessed via health record review and self-report (in the event of inconsistency, objective data will dominate).
Self-reported days of opioid use in the past 30 days | Baseline to 3-, 6-, and 12-months
  Self-reported days of non-prescribed opioid use in the past 30 days will be assessed at each interview.
Opioid use | 3-, 6-, and 12-month follow-up
  Positive oral fluid test for non-prescribed opioids (e.g., fentanyl, heroin, etc.)
Overdose events | through 3, 6, and 12 months
  Overdose events will be assessed by self-report and health records (for non-fatal events) and death records (for fatal events)
Changes in Social Support from Baseline to Follow-up | Baseline to 3-, 6-, and 12-month follow-up
  Social support will be measured using the Social Support Scale to determine the extent to which services influenced social support. It is a numeric scale from 0 to 100, with higher scores indicating greater social support.
Changes in Quality of Life from Baseline to Follow-up | Baseline to 3-, 6-, and 12-month follow up
  Quality of life will be measured via the World Health Organization Quality of Life instrument. It is a numeric scale with scores possible from 4-20, with higher scores indicating higher quality of life.
Changes in Psychological distress from baseline | Baseline to 3-, 6- and 12-month follow-up
  Kessler Psychological Distress Scale will be used to assess how participants have been feeling (nervous, hopeless, restless, depressed, worthless, etc) during their last 30 days. It is a numeric scale with scores ranging from 0 to 24, with higher scores indicating greater psychological distress.

OTHER OUTCOMES:
Rate of Patient-Directed Discharge | At discharge (assessed up to 12 months)
  Patient-directed discharge from the index hospitalization (i.e., "against medical advice") will be determined by health record review.
Mortality | through 12 months
  Mortality will be tracked from participant monitoring and death records

CONTACTS AND LOCATIONS:
Locations (1):
- Jefferson Health, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will complete baseline surveys and follow-up study surveys, and some participants will complete qualitative interviews. The raw interview and survey data will be stored within a secure computing environment. Metadata, study protocols, data collection instruments (surveys, interview guides), codebooks, and de-identified versions of participant data will be preserved and shared as appropriate to facilitate interpretation and reuse.
Supporting Information: Study Protocol
Time Frame: De-identified data and metadata will be deposited in a recognized repository such as the Inter-university Consortium for Political and Social Research (ICPSR) or another NIH-approved repository recommended by NINR. Once archived, datasets will be assigned persistent unique identifiers (such as DOIs) and indexed using repository tools and NIH-mandated descriptors to ensure they are findable and citable.
  De-identified data will be made available no later than the first publication of primary results or the end of the performance period, whichever comes first. Derived or summary datasets associated with publications will be shared with minimal delay. Shared data will remain available for at least five years following project completion, or longer if required by the repository or by NIH policy.
Access Criteria: FRI is committed to facilitating access to study data for individual researchers or other stakeholders, upon reasonable request and execution of a data sharing and use agreement

REFERENCES:
- [Background] Gryczynski J, Nordeck CD, Welsh C, Mitchell SG, O'Grady KE, Schwartz RP. Preventing Hospital Readmission for Patients With Comorbid Substance Use Disorder : A Randomized Trial. Ann Intern Med. 2021 Jul;174(7):899-909. doi: 10.7326/M20-5475. Epub 2021 Apr 6. PMID 33819055